CLINICAL TRIAL: NCT03212313
Title: A Two-Part, Open-Label, Single-Dose Study to Investigate the Influence of Hepatic Insufficiency on the Pharmacokinetics of Tozadenant
Brief Title: Study to Investigate the Influence of Hepatic Insufficiency on the Pharmacokinetics of Tozadenant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New Safety Information
Sponsor: Biotie Therapies Inc. (Industry)
Collaborators: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: TOZ-CL11
Record Dates: First submitted 2017-06-30; First posted 2017-07-11 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-07

CONDITIONS: Hepatic Impairment
Keywords: Adults; Liver Disease
MeSH Terms: conditions — Liver Diseases | interventions — tozadenant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy Subjects (Active Comparator): Study dose of 120 mg
  Interventions: Drug: Tozadenant
- Mild Hepatic Impairment (Experimental): Study dose of 120 mg
  Interventions: Drug: Tozadenant
- Moderate Hepatic Impairment (Experimental): Study dose of 120 mg
  Interventions: Drug: Tozadenant
- Severe Hepatic Impairment (Experimental): Up to a maximum study dose of 120 mg
  Interventions: Drug: Tozadenant

INTERVENTIONS:
Drug: Tozadenant — Two 60 mg tablets for a total single study dose of 120 mg

SUMMARY:
This is a two-part, open label, single-dose study that will evaluate the PK of tozadenant in subjects with different degrees of hepatic impairment to the PK of a single-dose of tozadenant in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

All subjects must fulfill the following to participate:

* Subject has given his/her written informed consent on an IEC or IRB approved consent form.
* Subject understands the study procedures in the informed consent form (ICF), and is willing and able to comply with the protocol.
* Be either male or female 18 years old
* Have a BMI ≥ 18.5 and ≤ 40.0 kg/m2 at screening
* Is a continuous non-smoker or a smoker who will consume up to 10 cigarettes/day
* Child bearing females should be sexually inactive (abstinent) prior to dosing
* Females subjects of non childbearing potential must have undergone one of the following sterilization or be postmenopausal

Subjects with mild, moderate, or severe hepatic impairment must:

* Have a medical history consistent with a diagnosis of hepatic impairment.
* Have a diagnosis of chronic (> 6 months), stable hepatic insufficiency

Healthy subjects must be:

* Medically healthy with no significant medical history

Exclusion Criteria:

Subjects must not be enrolled in the study if they:

* Previously participated in any study with tozadenant
* Has orthostatic hypotension, history or symptoms of cardiovascular disease, or hypertensive crisis.
* Currently participating in or has participated in another study and received drug (active or placebo)
* Have a known diagnosis of malignant melanoma
* Have a current episode of major depression
* Has a recent history of suicide attempt
* Has any other condition or clinically significant abnormal findings on the physical or neurological examination, psychiatric and medical history
* Had surgery or any medical condition within 6 months
* Unable to refrain from or anticipates the use of any drugs, vitamins, natural or herbal supplements
* Subject is currently lactating or pregnant or planning to become pregnant.
* Recent donation of blood, plasma or significant blood loss
* Has positive test for ethanol or drugs of abuse or a history of chronic alcohol or drug abuse
* Clinically significant medical history
* Positive results hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) for Healthy Volunteers only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics (PK) [area under the time-concentration curve] of a single-dose of tozadenant in subjects with hepatic impairment to healthy subjects. | up to 12 days
  To evaluate the pharmacokinetics (PK) [area under the time-concentration curve] of a single-dose of tozadenant in subjects with hepatic impairment compared to the PK of a single-dose of tozadenant in healthy subjects.

SECONDARY OUTCOMES:
Subjects with hepatic impairment will be evaluated for safety assessments (adverse events and treatment-related adverse events) by physical examinations. | up to 12 days
  To evaluate the safety and tolerability of a single-dose of tozadenant in subjects with hepatic impairment by physical examinations, vital sign measurements and Columbia-Suicide Severity Rating Scale (C-SSRS) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Preston, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No